CLINICAL TRIAL: NCT01437488
Title: A Phase II Study of Cabazitaxel in Patients With Urothelial Carcinoma Who Have Disease Progression Following Platinum-Based Chemotherapy
Brief Title: Cabazitaxel in Patients With Urothelial Carcinoma Who Have Disease Progression Following Platinum-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11D.392; 2011-52 (Other: CCRRC); JT 2205 (Other: JeffTrial Number)
Record Dates: First submitted 2011-08-31; First posted 2011-09-21 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial carcinoma; Urothelial cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — cabazitaxel; XRP6258; pegfilgrastim; Tomography Scanners, X-Ray Computed; Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (Experimental): Cabazitaxel following platinum-based chemotherapy
  Interventions: Drug: Cabazitaxel; Drug: Neulasta; Procedure: CT Scan; Biological: Blood Draw

INTERVENTIONS:
Drug: Cabazitaxel — * Cycle 1: 20 mg/m2 in 250cc NS via IV on Day 1 every 21 days
  * Following cycles: 20 mg/m2 or escalated to 25 mg/m2 or reduced by 5 mg/m2 in 250cc NS via IV on Day 1 every 21 days at investigator's discretion
  * Treatment continues until disease progression, intercurrent illness preventing further treatment, unacceptable adverse event(s), patient withdraws from the study, or changes in the patient's condition which render further treatment unacceptable in the judgment of the investigator
  Other Names: XRP-6258; Jevtana
Drug: Neulasta — 6 mg via SQ on Day 2 (24-48 hours post-cabazitaxel) every 21 days
  Other Names: Pegfilgrastim
Procedure: CT Scan — CT scan of chest, abdomen, and pelvis to assess disease following every 3rd cycle of treatment (approximately every 9 weeks)
  Other Names: X-ray computed tomography
Biological: Blood Draw — Approximately 2 tablespoons of blood will be taken to test complete blood count, glucose, hematology, electrolytes, liver function, creatinine clearance, and a chemistry profile. This week be done weekly during the first cycle of treatment
  Other Names: Venipuncture

SUMMARY:
There is no accepted standard chemotherapy approved for use in the second line for patients with advanced urothelial carcinoma whose cancer has progressed on combination chemotherapy including either cisplatin or carboplatin. The chemotherapy class called taxanes, either as single agents or in combination, have demonstrated modest efficacy in small studies. Cabazitaxel is an agent in the taxane family designed to be active in the setting of acquired multi-drug resistance that arises in some tumors. The objective of this study is to evaluate the safety and efficacy of this agent in patients with urothelial carcinoma refractory compared to combination platinum based chemotherapy.

DETAILED DESCRIPTION:
This is a single-arm, open-label study, meaning all patients will be treated in the same fashion with the investigational agent. Scans will be performed every 3 cycles of treatment, and patients will be withdrawn from study in the event of progression or drug intolerance as defined within the protocol.

Treatment will be administered on an outpatient basis. No investigational or commercial agents or therapies other than those described below may be administered with the intent to treat the patient's malignancy.

The length of each cycle is 21 days. For the first cycle of treatment, cabazitaxel will be dosed at 20 mg/m2. During cycle 1, complete blood counts will be performed on days 8 and 15, and dosing on Day 1 cycle 2 will depend upon the nadir counts on those days. If, on toxicity assessment on day 1 of cycle 2, the patient has no residual >grade 2 toxicity, and all other laboratory parameters are within acceptable limits (see below),at the investigator's discretion the dose can be escalated to 25 mg/m2. 25 mg/m2 is the FDA (Food and Drug Administration)-approved dose for prostate cancer. Neulasta will be given with each dose of cabazitaxel to decrease the risk of febrile neutropenic complication.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed urothelial carcinoma
* Patients must have measurable disease
* Patients must have been previously treated with a platinum-based regimen, either in the neoadjuvant, adjuvant or first line setting
* Patients can have had disease progression while on platinum chemotherapy, or progression within 12 months of completion of therapy
* At least 4 weeks must have passed since the last dose of previous chemotherapy
* Age > 18 years
* ECOG performance status < 2 (Karnofsky > 60%)
* Life expectancy of greater than 6 months
* Patients must have adequate organ and marrow function as defined below:
* absolute neutrophil count > 1,500/mcL
* hemoglobin > 9.0 g/dl
* platelets > 100,000/mm3
* total bilirubin < normal institutional limits (ULN)
* AST(SGOT)/ALT(SGPT) < 1.5 X institutional upper limit of normal
* creatinine <1.5 x ULN OR creatinine clearance measured > 50 mL/min/1.73 m2for patients with creatinine levels above institutional normal or calculated clearance < 60 by 24 hour urine
* Peripheral neuropathy: must be < grade 1
* Women of childbearing potential must have a negative pregnancy test, and patients must use adequate contraception during study and for 3 months thereafter
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with any component of small cell carcinoma
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to taxane chemotherapy
* Patients with a history of severe hypersensitivity reaction to Cabazitaxel or other drugs formulated with polysorbate 80
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and breastfeeding women
* HIV-positive patients on combination antiretroviral therapy
* Patients who have previously been treated with taxane regimens for bladder cancer or other malignancies
* Patients who have had more than one platinum based chemotherapy regimen
* Patients whose cancer has progressed more than 12 months following abstinence from platinum based chemotherapy can be included on study at the discretion of the investigator, however should first be considered for platinum re-challenge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02-16 (Actual); Primary Completion 2014-08-04 (Actual); Study Completion 2017-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Hoffman-Censits, MD, Principal Investigator — Thomas Jefferson University
Locations (3):
- United States (3):
  - National Cancer Institute, Bethesda, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://www.jeffersonhospital.org/
- See also: Center for Cancer Research, National Cancer Institute — http://ccr.cancer.gov/
- See also: Abramson Cancer Center of the University of Pennsylvania — http://penncancer.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cabazitaxel: Cabazitaxel following platinum-based chemotherapy Cabazitaxel: - Cycle 1: 20 mg/m2 in 250cc NS via IV on Day 1 every 21 days
  * Following cycles: 20 mg/m2 or escalated to 25 mg/m2 or reduced by 5 mg/m2 in 250cc NS via IV on Day 1 every 21 days at investigator's discretion
  * Treatment continues until disease progression, intercurrent illness preventing further treatment, unacceptable adverse event(s), patient withdraws from the study, or changes in the patient's condition which render further treatment unacceptable in the judgment of the investigator
  Neulasta: 6 mg via SQ on Day 2 (24-48 hours post-cabazitaxel) every 21 days
  CT Scan: CT scan of chest, abdomen, and pelvis to assess disease following every 3rd cycle of treatment (approximately every 9 weeks)
  Blood Draw: Approximately 2 tablespoons of blood will be taken to test complete blood count, glucose, hematology, electrolytes, liver function, creatinine clearance, and a chemistry profile. This week be done weekly durin
Period: Overall Study
Arm/Group | Cabazitaxel
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cabazitaxel
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To determine the overall response rate of patients who have disease response while on treatment with Cabazitaxel. CT scan will be used to measure tumor pre-treatment and then every 3 cycles (every 63 days)
Time Frame: Every 3 cycles or 63 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cabazitaxel
Number analyzed (Participants) | 14
Participants | 11

2. Secondary Outcome: Overall Survival
Description: To determine the percentage of patients alive at 12 months from trial entry. Overall survival will be measured from date of randomization to date of death due to any cause.
Time Frame: At 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Cabazitaxel: Cabazitaxel: - Cycle 1: 20 mg/m2 in 250cc NS via IV on Day 1 every 21 days
  * Following cycles: 20 mg/m2 or escalated to 25 mg/m2 or reduced by 5 mg/m2 in 250cc NS via IV on Day 1 every 21 days at investigator's discretion
  * Treatment continues until disease progression, intercurrent illness preventing further treatment, unacceptable adverse event(s), patient withdraws from the study, or changes in the patient's condition which render further treatment unacceptable in the judgment of the investigator Neulasta: 6 mg via SQ on Day 2 (24-48 hours post-cabazitaxel) every 21 days CT Scan: CT scan of chest, abdomen, and pelvis to assess disease following every 3rd cycle of treatment (approximately every 9 weeks) Blood Draw: Approximately 2 tablespoons of blood will be taken to test complete blood count, glucose, hematology, electrolytes, liver function, creatinine clearance, and a chemistry profile. This week be done weekly during the first cycle of treatment
Arm/Group | Cabazitaxel
Number analyzed (Participants) | 14
Participants | 13

3. Secondary Outcome: Progression Free Survival
Description: To determine the progression free survival (PFS) of patients with advanced or recurrent urothelial carcinoma who have previously been treated with a platinum based regimen while on treatment with cabazitaxel. Defined as a 20% increase in the largest diameter of the largest lesion by CT scan.
Time Frame: Every 3 cycles or 63 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cabazitaxel
Number analyzed (Participants) | 14
Participants | 11

4. Secondary Outcome: Number of Participants Who Tolerated Cabazitaxel
Time Frame: Up to 30 days after completion of study treatment
Measure: Count of Participants; unit: Participants
Groups:
- Cabazitaxel: Cabazitaxel following platinum-based chemotherapy
  Cabazitaxel: - Cycle 1: 20 mg/m2 in 250cc NS via IV on Day 1 every 21 days
  * Following cycles: 20 mg/m2 or escalated to 25 mg/m2 or reduced by 5 mg/m2 in 250cc NS via IV on Day 1 every 21 days at investigator's discretion
  * Treatment continues until disease progression, intercurrent illness preventing further treatment, unacceptable adverse event(s), patient withdraws from the study, or changes in the patient's condition which render further treatment unacceptable in the judgment of the investigator
  Neulasta: 6 mg via SQ on Day 2 (24-48 hours post-cabazitaxel) every 21 days
  CT Scan: CT scan of chest, abdomen, and pelvis to assess disease following every 3rd cycle of treatment (approximately every 9 weeks)
  Blood Draw: Approximately 2 tablespoons of blood will be taken to test complete blood count, glucose, hematology, electrolytes, liver function, creatinine clearance, and a chemistry profile.
Arm/Group | Cabazitaxel
Number analyzed (Participants) | 14
Participants | 11

ADVERSE EVENTS:
Time Frame: Every 21 days, up to 1 year
Arm/Group | Cabazitaxel
All-Cause Mortality (participants affected / at risk) | 1/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabazitaxel (N=14)
Embolic stroke (Blood and lymphatic system disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabazitaxel (N=14)
Fatigue (General disorders) | 9 (10)
Abdominal cramping (Musculoskeletal and connective tissue disorders) | 2 (2)
Abdominal distention (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Acid Reflux (Gastrointestinal disorders) | 1 (1)
Alkalosis (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Anorexia (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder Spasm (Renal and urinary disorders) | 1 (1)
Bleeding Gums (General disorders) | 1 (1)
Bloating (General disorders) | 1 (1)
Blood in Bilirubin increased (Blood and lymphatic system disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cabazitaxel Infusion reaction (Product Issues) | 1 (1)
Change in Taste (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Creatinine Increased (Blood and lymphatic system disorders) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dizziness (Nervous system disorders) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Epigastric Pain (Gastrointestinal disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Fever (Infections and infestations) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu-Like symptoms (Infections and infestations) | 2 (2)
Foot Pain (General disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hematuria (Blood and lymphatic system disorders) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 3 (3)
Hypomagnesia (Blood and lymphatic system disorders) | 2 (2)
INR increased (Blood and lymphatic system disorders) | 1 (1)
Insomnia (Nervous system disorders) | 2 (2)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lightheadedness (General disorders) | 3 (3)
Loose Stools (Gastrointestinal disorders) | 1 (1)
mild-mod Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (6)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Pain in Pelvis (General disorders) | 1 (1)
Paresthesia bilateral feet (Nervous system disorders) | 1 (1)
Perioral numbness (Nervous system disorders) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 1 (2)
Pinching sensation around port (General disorders) | 2 (2)
PTT prolonged (General disorders) | 1 (2)
Pyelonephritis (Hepatobiliary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rib pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sacral Edema (General disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Tearing (Eye disorders) | 1 (1)
Throat discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Tinnitus (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
URI (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Vision changes (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Worsening pain (General disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes